CLINICAL TRIAL: NCT00786734
Title: A Randomized, Open Label, Comparative Study to Evaluate Effect of Pitavastatin for Reduction of Myocardial Damage in Patient Are Scheduled Elective PCI for Stable Angina Pectoris
Brief Title: Pitavastatin Pre-Treatment Study in Patient With Elective PCI for Stable Angina Pectoris (PIPA)
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CWP-PTV-705
Record Dates: First submitted 2008-11-05; First posted 2008-11-06 (Estimated); Last update posted 2012-03-30 (Estimated); Status verified 2012-03

CONDITIONS: Percutaneous Coronary Intervention
Keywords: pitavastatin; PCI; stable angina
MeSH Terms: conditions — Angina, Stable | interventions — pitavastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pitavastatin Group (Experimental)
  Interventions: Drug: Pitavastatin
- Usual Care Group (Other)
  Interventions: Drug: Pitavastatin

INTERVENTIONS:
Drug: Pitavastatin — 4mg daily for 5-7 days before Percutaneous Coronary Intervention(PCI) and 4mg daily for 28 days after PCI
  Arms: Pitavastatin Group
Drug: Pitavastatin — 4mg daily for 28 days after PCI
  Arms: Usual Care Group

SUMMARY:
Patients who is scheduled elective PCI are randomized to pitavastatin 4mg daily or without pitavastatin for 5 -7days before the procedure. Creatine kinase-MB, troponin I, and myoglobin levels are measured at baseline and at 8 and 24 hours after the procedure(1st evaluation). After PCI, pitavastatin will be administered for additional 4 weeks(2nd evaluation).

DETAILED DESCRIPTION:
Procedural ischemic myocardial injury remains the most frequent complication after coronary angioplasty. Recently it was reported that pretreatment with atorvastatin reduce the myocardial damage compared to placebo. Thus, we will evaluate the difference of pretreatment of pitavastatin compared to standard therapy on the reduction of myocardial damage in patient who is scheduled elective PCI for stable angina pectoris.

ELIGIBILITY:
Inclusion Criteria:

* Patients with LDL ≥ 100mg/dL
* Patients who are scheduled an elective PCI for stable angina

Exclusion Criteria:

* Acute myocardial infarction (<3 months)
* Unstable angina
* Previous treatment with statins (<6 months)
* Increase in CK-MB above upper normal limit
* Increase in liver enzymes (AST/ALT) above 2 times of upper normal limit
* Increase in serum creatinine above 2 times of upper normal limit
* Left ventricular ejection fraction <30%
* Previous treatment with glycoprotein Ⅱb/Ⅲa receptor inhibitor (<4 weeks)

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-08; Primary Completion 2009-05 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Proportion of patients whose CK-MB > 2 times above UNL | First evaulation time (before PCI)

SECONDARY OUTCOMES:
Proportion of patients who show any increase of CK-MB, troponin I, and myoglobin above UNL | First evaluation time
Mean peak values of CK-MB, troponin I and myoglobin after intervention | After PCI (<24hrs)
Change of hs-CRP, wall motion score | Second evaluation time
Occurence of all major adverse cardiac events | Second evaluation time

CONTACTS AND LOCATIONS:
Overall Officials: Ki Bae Seung, Ph.D, Principal Investigator — Professor, Catholic University of Korea Kangnam St. Mary's Hospital located
Locations (1):
- Catholic University of Korea Kangnam St. Mary's Hospital, Seoul, South Korea